CLINICAL TRIAL: NCT05702983
Title: An Open-label, Single-ascending Dose, Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of STSA-1002 Subcutaneous Injection in Healthy Subjects
Brief Title: The Safety and Tolerability of STSA-1002 Following Subcutaneous Injection in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STSA-1002-S01
Record Dates: First submitted 2022-12-23; First posted 2023-01-27 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Antineutrophil Cytoplasmic Antibody Associated Vasculitis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- STSA-1002 subcutaneous injection: dose 1 (First cohort) (Experimental)
  Interventions: Drug: STSA-1002 subcutaneous injection
- STSA-1002 subcutaneous injection: dose 2 (Second cohort) (Experimental)
  Interventions: Drug: STSA-1002 subcutaneous injection

INTERVENTIONS:
Drug: STSA-1002 subcutaneous injection — Subjects will receive a single low dose on day 1 following protocol requirements.
  Arms: STSA-1002 subcutaneous injection: dose 1 (First cohort)
Drug: STSA-1002 subcutaneous injection — Subjects will receive a single high dose on day 1 following protocol requirements.
  Arms: STSA-1002 subcutaneous injection: dose 2 (Second cohort)

SUMMARY:
An Open-label, Single-ascending dose, Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of STSA-1002 Subcutaneous Injection in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, aged ≥ 21 but ≤ 57, male and female.
* Weight: 50-93 kg; Body mass index (BMI): 21～31 kg/m2, inclusive.
* Subjects (including their partners) agree to take highly effective contraceptive measures during the study, and they have no birth plan or sperm donation plan within 6 months after the end of the study.
* Female and/or male subjects those meet the below criteria:

If a female subject of childbearing potential - agrees to use one of the accepted contraceptive regimens from at least 30 days prior to administration of IMP, during the study, and for at least 6 months after the administration of IMP. An acceptable method of contraception includes one of the following:

Abstinence from heterosexual intercourse, if it is the preferred and usual lifestyle choice of the subject. Additionally, it should be noted that periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) is not an acceptable method of birth control; Hormonal contraceptives (birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch); Intrauterine device (with or without hormones) OR agrees to use a double barrier method (e.g. condom and spermicide) during the study and for at 6 months after the administration of IMP.

If a female subject of non-childbearing potential - should have been surgically sterilized at least 6 months before screening (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation/occlusion) or in the postmenopausal state (at least 1 year without menses), as confirmed by Follicle-stimulating hormone (FSH) levels (≥ 40 mIU/mL).

A male subject that engages in sexual activity that has the risk of pregnancy must agree to use a double barrier method (e.g. condom and spermicide) and agree to not donate sperm during the study and for at least 6 months after the administration of IMP.

* Medical histories, physical examinations, laboratory examinations and study-related examinations and tests of the subjects show normal results or mild abnormalities with no clinical significance before enrollment, and the Investigator judges that they are eligible.
* Subjects are aware of the risks of the study, and voluntarily participate in the clinical study and sign an informed consent form (ICF).

Exclusion Criteria:

* History of cardiovascular, respiratory, kidney, liver, metabolism, endocrine, gastrointestinal, blood, nerve, skin and mental illness, cancer or other major disease that in the judgment of the Investigator might put the subject as risk on this study.
* History of tuberculosis or a recent history of infection within the past 4 weeks.
* History of recurrent infections.
* Presence of clinically significant laboratory values during the screening period, as defined by an Investigator.
* Presence of clinically significant vital signs values or of electrocardiogram (ECG) abnormalities during the screening period, as defined by an Investigator.
* Subjects who have autoimmune disease or immunodeficiency, or have a family history of related diseases.
* Subjects who have history of hypersensitivity or clinically significant allergic reaction to any drug, biologic, food or vaccine.
* Positive screening test results for human immunodeficiency virus (HIV-1/HIV-2) antibodies, hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCVAb).
* Subjects who have received treatment with an investigational drug within 30 days or 5 times the half-life (whichever is longer) prior to screening.
* Subjects who have participated in any vaccine clinical study or have received any live vaccine within 3 months prior to the IMP administration or plan to receive live vaccines during the study period, and subjects who have received inactivated or attenuated vaccines 28 days prior to the IMP administration or plan to receive inactivated or attenuated vaccines within 2 months after the end of the study. If the subject has received any SARS-CoV-2 vaccine prior to screening, enrollment must be delayed until the biologic impact of the vaccine is stabilized, as determined by discussion between the investigator and the sponsor.
* Subjects who have taken drugs that may affect immune function within 6 months before screening, have received any monoclonal antibody or biological agent for treatment (for any illness) within the previous 3 months, and have previous treatment with any prescribed medications (including vaccines) or over-the-counter (OTC) medications (including herbal medicines such as St John's Wort, homeopathic preparations, vitamins, and minerals) within 7 days prior to IMP administration.
* Subjects whose daily consumption of coffee, tea and/or cola is more than 750 mL or 25 fl. oz in the last 30 days before enrollment.
* Subjects who have a positive urine alcohol test or urine drug test before enrollment.
* Subjects who have nicotine consumption (e.g., smoking, nicotine patch, nicotine chewing gum, or electronic cigarettes) within 3 months prior to screening and inability to refrain from nicotine consumption from screening until end of study.
* Female subjects who are pregnant or breastfeeding during the screening period and on admission.
* Subjects whose daily consumption of alcohol at the time of screening or at any time within the prior 2 months is more than 2 standard drinks, where 1 standard drink = 355 mL or 12 oz (1 can) of regular-strength (5%) beer; 150 mL or 5 oz wine; 45 mL or 1.5 oz liquor/spirits (40%).
* History of drug or alcohol abuse (as defined by the investigator), or addiction within 1 year prior to screening.
* Subjects who have undergone major surgery within 6 months of screening, or who will have elective surgery that will occur during the study period.
* Subjects who have donated either more than approximately 500 mL of blood (exclusive plasma donation) within 56 days (8 weeks) prior to screening or any plasma within 7 days (1 week) prior to screening.
* Subjects fails or is unwilling to abstain from strenuous physical activities for at least 48 hours prior to IMP administration and throughout the study.
* Subjects with any factors that would, in the Investigator's judgment, preclude them from participating in this study.

Ages: 21 Years to 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Number of treatment-related adverse events as assessed by toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials | 50 days
  To evaluate the safety and tolerability of STSA-1002 subcutaneous injection in healthy adult subjects
Abnormal clinical laboratory values as assessed by toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials (blood hematology, blood chemistry, urinalysis, etc.) | 50 days
  To evaluate the safety and tolerability of STSA-1002 subcutaneous injection in healthy adult subjects
Abnormal vital signs as assessed by toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials (body temperature, pulse rate, blood pressure and respiratory rate) | 50 days
  To evaluate the safety and tolerability of STSA-1002 subcutaneous injection in healthy adult subjects
Abnormal physical examination | 50 days
  To evaluate the safety and tolerability of STSA-1002 subcutaneous injection in healthy adult subjects
Abnormal electrocardiogram (ECG): heart rate, PR and QT intervals, QTcF and QRS duration | 50 days
  To evaluate the safety and tolerability of STSA-1002 subcutaneous injection in healthy adult subjects
Maximum plasma concentration (Cmax) | Pre-dose; after dose 8hours, 24hours, 48hours, 72hours, 96hours, 120hours, 168hours, 336hours, 504hours, 840hours, 1176hours
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1002 subcutaneous injection in healthy adult subjects
area under the plasma concentration-time curve from time 0 to the collection time point t of the last measurable concentration (AUC0-t) | Pre-dose; after dose 8hours, 24hours, 48hours, 72hours, 96hours, 120hours, 168hours, 336hours, 504hours, 840hours, 1176hours
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1002 subcutaneous injection in healthy adult subjects
area under the plasma concentration-time curve from time 0 to infinity (AUC0-∞) | Pre-dose; after dose 8hours, 24hours, 48hours, 72hours, 96hours, 120hours, 168hours, 336hours, 504hours, 840hours, 1176hours
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1002 subcutaneous injection in healthy adult subjects
Time of maximum concentration (Tmax) | Pre-dose; after dose 8hours, 24hours, 48hours, 72hours, 96hours, 120hours, 168hours, 336hours, 504hours, 840hours, 1176hours
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1002 subcutaneous injection in healthy adult subjects
elimination half-life (t1/2) | Pre-dose; after dose 8hours, 24hours, 48hours, 72hours, 96hours, 120hours, 168hours, 336hours, 504hours, 840hours, 1176hours
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1002 subcutaneous injection in healthy adult subjects
elimination rate constant of plasma drug concentration in terminal phase (λz) | Pre-dose; after dose 8hours, 24hours, 48hours, 72hours, 96hours, 120hours, 168hours, 336hours, 504hours, 840hours, 1176hours
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1002 subcutaneous injection in healthy adult subjects
last measurable concentration (Clast) | Pre-dose; after dose 8hours, 24hours, 48hours, 72hours, 96hours, 120hours, 168hours, 336hours, 504hours, 840hours, 1176hours
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1002 subcutaneous injection in healthy adult subjects
mean residence time (MRT) | Pre-dose; after dose 8hours, 24hours, 48hours, 72hours, 96hours, 120hours, 168hours, 336hours, 504hours, 840hours, 1176hours
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1002 subcutaneous injection in healthy adult subjects
clearance (CL) | Pre-dose; after dose 8hours, 24hours, 48hours, 72hours, 96hours, 120hours, 168hours, 336hours, 504hours, 840hours, 1176hours
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1002 subcutaneous injection in healthy adult subjects
apparent volume of distribution (Vz) | Pre-dose; after dose 8hours, 24hours, 48hours, 72hours, 96hours, 120hours, 168hours, 336hours, 504hours, 840hours, 1176hours
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1002 subcutaneous injection in healthy adult subjects

SECONDARY OUTCOMES:
Change from baseline in concentration of free C5a | Pre-dose; after dose 8hours, 24hours, 48hours, 72hours, 96hours, 120hours, 168hours, 336hours, 504hours, 840hours, 1176hours
  To evaluate the pharmacodynamics (PD) characteristics and immunogenicity of STSA-1002 subcutaneous injection in healthy subjects
anti-drug antibody | Pre-dose; after dose 336hours, 840hours, 1176hours
  To evaluate the pharmacodynamics (PD) characteristics and immunogenicity of STSA-1002 subcutaneous injection in healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Martin K Kankam, Doctor, Principal Investigator — Altasciences Clinical Kansas, Inc.
Locations (1):
- AltaSciences Clinical Kansas, Inc, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No